CLINICAL TRIAL: NCT01232127
Title: Open-Label, Multiple-Dose, Drug Interaction Study to Assess the Effect of Famotidine on the Pharmacokinetics of Atazanavir in HIV-Infected Subjects Receiving Atazanavir With Ritonavir and Tenofovir
Brief Title: Effects of Famotidine on the Pharmacokinetics of Atazanavir When Coadministered to Participants With HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AI424-398; 2009-016981-95 (EudraCT Number)
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: HIV
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir; Tenofovir; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atazanavir/ritonavir (300/100 mg) + TDF + ≥ 1 NRTI (Other): The protocol required that participants enrolled in this study already be receiving atazanavir, ritonavir, TDF, and 1 or more NRTIs.
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Tenofovir (TDF); Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTI)
- Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (20) (Other): FAM=famotidine. The protocol required that participants enrolled in this study already be receiving atazanavir, ritonavir, TDF, and 1 or more NRTIs.
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Tenofovir (TDF); Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTI); Drug: Famotidine (FAM)
- Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (40) (Other): FAM=famotidine. The protocol required that participants enrolled in this study already be receiving atazanavir, ritonavir, TDF, and 1 or more NRTIs.
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Tenofovir (TDF); Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTI); Drug: Famotidine (FAM)

INTERVENTIONS:
Drug: Atazanavir — Capsule, oral, 300 mg, once daily, 10 days
  Other Names: Reyataz; BMS-232632
  Arms: Atazanavir/ritonavir (300/100 mg) + TDF + ≥ 1 NRTI
Drug: Atazanavir — Capsule, oral, 400 mg, once daily, 7 days
  Other Names: Reyataz; BMS-232632
  Arms: Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (20); Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (40)
Drug: Ritonavir — Capsule, oral, 100 mg, once daily, 10 days
  Arms: Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (20); Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (40)
Drug: Ritonavir — Capsule, oral, 100 mg, once daily, 7 days
  Arms: Atazanavir/ritonavir (300/100 mg) + TDF + ≥ 1 NRTI
Drug: Tenofovir (TDF) — Capsule, oral, 300 mg, once daily, 10 days
  Arms: Atazanavir/ritonavir (300/100 mg) + TDF + ≥ 1 NRTI
Drug: Tenofovir (TDF) — Capsule, oral, 300 mg, once daily, 7 days
  Arms: Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (20); Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (40)
Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTI) — Oral, 10 days
  Arms: Atazanavir/ritonavir (300/100 mg) + TDF + ≥ 1 NRTI
Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTI) — Oral, 7 days
  Arms: Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (20); Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (40)
Drug: Famotidine (FAM) — Tablet, oral, 20 mg, twice daily, 7 days
  Arms: Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (20)
Drug: Famotidine (FAM) — Tablet, oral, 40 mg, twice daily, 7 days
  Arms: Atazanavir/ritonavir (400/100) + TDF + ≥1 NRTI + FAM (40)

SUMMARY:
The purpose of this study is to assess the effects of famotidine, given twice daily, on atazanavir administered with ritonavir and tenofovir in HIV-infected participants.

DETAILED DESCRIPTION:
This protocol was designed to compare the pharmacokinetic parameters of atazanavir administered as atazanavir/ritonavir, 400/100 mg once daily (QD), plus famotidine, 20 mg and 40 mg twice daily, with the parameters found at the usual clinical dose of atazanavir/ritonavir, 300/100 mg QD, without famotidine in HIV-infected participants receiving tenofovir disoproxil fumarate and at least 1 other nucleoside reverse transcriptase inhibitor.

ELIGIBILITY:
Key inclusion criteria:

* Males and females, 18 to 65 years of age, with HIV infection and a body mass index of 18.0 to 35.0 kg/m^2
* HIV-infected participants receiving a treatment regimen containing only atazanavir/ritonavir, 300/100 mg once daily (QD) + tenofovir, 300 mg QD + at least 1 other nucleotide reverse transcriptase inhibitor continuously for at least 3 months prior to study day 1
* Plasma HIV RNA levels of <50 copies/mL and a CD4 count >200 cells/mm^3.
* No history of virologic failure on a protease inhibitor (PI), documented phenotypic PI resistance, or primary PI mutations, according to International AIDS Society recommendations
* No documented phenotypic resistance to atazanavir or primary genotypic mutations causing resistance to atazanavir
* Women of childbearing potential who were not nursing or pregnant and were using an acceptable method of contraception for at least 4 weeks before dosing, during the study, and for 8 weeks from the last dose of study drug.
* Women with a negative pregnancy test result within 24 hours prior to dosing with study medication
* Women not breastfeeding
* Men willing or able to agree to practice barrier contraception for the duration of the study and at least 3 months after dosing.

Key exclusion criteria:

* Any history of CD4 cell count <50 cells/mm^3
* Previously documented phenotypic or genotypic resistance to any of the currently prescribed NRTIs
* Any significant acute illness within 6 months of study day 1 or chronic medical illness unless stable or controlled by a nonprohibited medication
* Any major surgery within 4 weeks of study day 1
* Any gastrointestinal surgery that could impact upon the absorption of any study drug
* Inability to be venipunctured and/or tolerate venous access
* History of Gilbert's syndrome, hemophilia, chronic pancreatitis, hypochlorhydria, achlorhydria, clinically relevant gastroesophageal reflux disease, hiatal hernia, or peptic/gastric ulcer disease
* Intractable diarrhea (≥ 6 loose stools/day for at least 7 consecutive days) within 30 days prior to study day 1
* Recent (within 6 months prior to study day 1) drug or alcohol abuse
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, electrocardiogram (ECG)
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations, which would not be expected for the extent of HIV disease
* Any of the following on 12-lead ECG prior to dosing on study day 1, confirmed by repeat: PR ≥ 210 msec; QRS ≥ 120 msec; QT ≥ 500 msec; QTcF ≥ 450 msec
* Second- or third-degree A-V block or clinically relevant ECG abnormalities
* Positive urine screen for drugs of abuse at screening or prior to dosing without a valid prescription. Positive urine drug screen for cannabinoids with or without a prescription is not exclusionary
* Creatinine clearance, as estimated by method of Cockcroft and Gault, less than 60 mL/min
* Liver enzyme levels > 3* the upper limit of normal (ULN) prior to dosing on study day 1
* Total bilirubin level >10*ULN prior to study day 1
* Positive blood screen for hepatitis B surface antigen or hepatitis C antibody.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution, Berlin, Germany
- Local Institution, London, Greater London, United Kingdom

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI: Participants received atazanavir/ritonavir, 300/100 mg QD, plus tenofovir (TDF), 300 mg QD, and at least 1 nucleoside reverse transcriptase inhibitor (NRTI). Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
- Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20): Participants received atazanavir/ritonavir, 400/100 mg QD, plus TDF, 300 mg QD, plus at least 1 NRTI, plus famotidine, 20 mg BID. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
- Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40): Participants received atazanavir/ritonavir, 400/100 mg QD, plus TDF, 300 mg QD, plus at least 1 NRTI, plus famotidine, 40 mg BID. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
Period: Period 1: Days 1-10
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Started | 25 (Participants who received treatment.) | 0 | 0
Completed | 24 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Discontinued due to dosing error | 1 | 0 | 0
Period: Period 2: Days 11-17
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Started | 0 | 24 (Participants who received treatment.) | 0
Completed | 0 | 24 | 0
Not Completed | 0 | 0 | 0
Period: Period 3: Days 18-24
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Started | 0 | 0 | 24 (Participants who received treatment.)
Completed | 0 | 0 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Treated
Number analyzed (Participants) | 25
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 25
  65 years and older | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Age [Mean (Full Range); unit: Years] | 39.8 [23 to 62]
CD4 Absolute Count [Mean (Standard Deviation); unit: Cells/μL] — n=23 (n=evaluable participants)
  Cells/μL | 584.8 (194.09)
CD4 Percent of Total [Mean (Standard Deviation); unit: Percent of participants] — n=23 (n=evaluable participants)For 2 participants, baseline CD4 percent total and absolute count were performed as an unscheduled visit after the initial screening visit and thus, are not included in this summary.
  Percent of participants | 32.1 (7.10)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, AES, and AEs of Clinical Interest
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Days 1 through 25 (end of study), continuously, and at study discharge for those who discontinued prematurely.
Population: Participants who received study drug and were evaluable.
Measure: Number; unit: Participants
Groups:
- Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI: Participants received atazanavir/ritonavir, 300/100 mg QD, plus tenofovir (TDF), 300 mg QD, and at least 1 nucleoside reverse transcriptase inhibitor (NRTI) on Days 1 through 10. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
- Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20): Participants received atazanavir/ritonavir, 400/100 mg QD, plus TDF, 300 mg QD, plus at least 1 NRTI, plus famotidine, 20 mg BID on Days 11 through 17. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
- Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40): Participants received atazanavir/ritonavir, 400/100 mg QD, plus TDF, 300 mg QD, plus at least 1 NRTI, plus famotidine, 40 mg BID on Days 18 through 24. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Number analyzed (Participants) | 25 | 25 | 24
Participants
  Deaths | 0 | 0 | 0
  SAEs | 0 | 0 | 0
  AEs leading to discontinuation | 0 | 0 | 0
  AEs | 6 | 7 | 5
  AEs of clinical interest: Nausea | 0 | 2 | 0
  AEs of clinical interest: Diarrhea | 0 | 3 | 0

2. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Vital signs include temperature, respiratory rate, seated blood pressure, and heart rate.
Time Frame: Days 1, 11, 18, and 25 (end of study) and at study discharge for those who discontinued prematurely.
Population: Participants who received study drug and were evaluable.
Measure: Number; unit: Participants
Groups:
- All Treated: All participants who received at least 1 dose of atazanavir with ritonavir and tenofovir and with or without famotidine.
Arm/Group | All Treated
Number analyzed (Participants) | 25
Participants
  Isolated decrease in heart rate | 2
  Sporadic respiration rate >16 bpm | 11

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) and Trough Observed Plasma Concentration (Ctrough) for Atazanavir and Ritonavir
Time Frame: Days 10, 11, 17, 18, 24, and 25 (end of study) and at study discharge for those who discontinued prematurely.
Population: Participants who received study drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI: Participants received atazanavir/ritonavir, 300/100 mg once daily (QD), plus tenofovir (TDF), 300 mg QD, and at least 1 nucleoside reverse transcriptase inhibitor (NRTI)on Days 1 through 10. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
- Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20): Participants received atazanavir/ritonavir, 400/100 mg QD, plus TDF, 300 mg QD, plus at least 1 NRTI, plus famotidine, 20 mg twice daily (BID) on Days 11 through 17. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Number analyzed (Participants) | 25 | 24 | 24
ng/mL
  Atazanavir Cmax | 3512 (35.4) | 4131 (37.7) | 3322 (45.2)
  Atazanavir Ctrough | 496 (50.9) | 602 (60.3) | 494 (59.4)
  Ritonavir Cmax | 1141 (30.5) | 1148 (29.8) | 1096 (36.1)
  Ritonavir Ctrough | 45.8 (58.7) | 49.2 (66.8) | 47.3 (53.4)

4. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) for Atazanavir and Ritonavir
Time Frame: Days 10, 11, 17, 18, 24, and 25 (end of study) and at study discharge for those who discontinued prematurely.
Population: Participants who received study drug and had adequate PK profiles.
Measure: Median (Full Range); unit: Hours
Groups:
- Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI: Participants received atazanavir/ritonavir, 300/100 mg QD, plus TDF, 300 mg QD, and at least 1 NRTI on Days 1 through 10. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Number analyzed (Participants) | 25 | 24 | 24
Hours
  Atazanavir Tmax | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.10]
  Ritonavir Tmax | 4.0 [2.0 to 4.2] | 4.00 [2.0 to 6.0] | 4.0 [2.0 to 6.0]

5. Primary Outcome: Area Under the Plasma Concentration-time Curve in 1 Dosing Interval (Time 0 to 24 Hours Postdose) (AUC[TAU]) for Atazanavir and Ritonavir
Time Frame: Days 10, 11, 17, 18, 24, and 25 (end of study) and at study discharge for those who discontinued prematurely.
Population: Participants who received study drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Number analyzed (Participants) | 25 | 24 | 24
ng*h/mL
  Atazanavir AUC | 32562 (37.7) | 37894 (40.7) | 31481 (48.8)
  Ritonavir AUC | 7317 (35.6) | 7430 (32.4) | 7052 (36.7)

6. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiogram (ECG) Findings
Description: ECG findings include heart rate, ECG intervals (including PR, QRS, QT, and corrections to QT using both Bazett's and Fridericia's formulae), and Investigator-identified ECG abnormalities.
Time Frame: Days 1 and 25 (end of study) and at study discharge for those who discontinued prematurely.
Population: Participants who received study drug and were evaluable.
Measure: Number; unit: Participants
Arm/Group | All Treated
Number analyzed (Participants) | 25
Participants
  Nonspecific ST/T wave abnormality | 1
  Short PR interval | 1

7. Secondary Outcome: Number of Participants With Abnormalities in Laboratory Test Results
Description: PreRX=pretreatment; ULN=upper limit of normal. Neutrophils, (absolute), low (10*3 c/uL): <0.85*PreRx, if PreRx <1.5; <1.5 if PreRx ≥1.5. Alanine aminotransferase, high (U/L): >1.25*PreRx if PreRx >ULN; >1.25*ULN if PreRx ≤ULN. Bilirubin, direct (mg/dL), high: >1.1*ULN if PreRx ≤ULN;> 1.1*ULN if PreRx is missing; >1.25*PreRx if PreRx >ULN. Bilirubin, total (mg/dL), high: >1.1*ULN if PreRx ≤ULN;> 1.1*ULN if PreRx is missing; >1.25*PreRx if PreRx >ULN.
Time Frame: Days 11, 18, and 25 (end of study) and at study discharge for those who discontinued prematurely.
Population: Participants who received study drug and were evaluable.
Measure: Number; unit: Participants
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Number analyzed (Participants) | 25 | 24 | 23
Participants
  WBC differential count (low) | 1 | 0 | 0
  Neutrophils (absolute) (low) | 0 | 1 | 0
  Alanine aminotransferase (high) | 0 | 1 | 0
  Aspartate aminotransferase (high) | 0 | 0 | 1
  Bilirubin, direct (high) | 1 | 0 | 0
  Bilirubin, total (high) | 3 | 7 | 5

ADVERSE EVENTS:
Time Frame: Days 1 through 25 (end of study), continuously, and at study discharge for those who discontinued prematurely.
Groups:
- Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI: Participants received atazanavir/ritonavir, 300/100 mg once daily (QD), plus tenofovir (TDF), 300 mg QD, and at least 1 nucleoside reverse transcriptase inhibitor (NRTI) on Days 1 through 10. Atazanavir/ritonavir and TDF were administered with food. The AM dose of famotidine was administered simultaneously with atazanavir/ritonavir/TDF.
Arm/Group | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 4/25 | 6/25 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir/Ritonavir (300/100) + TDF + ≥NRTI (N=25) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (20) (N=25) | Atazanavir/Ritonavir (400/100) + TDF + ≥NRTI + Famotidine (40) (N=24)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.